CLINICAL TRIAL: NCT02027103
Title: Comparative Effects of Metformin and Pioglitazone on Fetuin-A and Osteoprotegerin Concentrations in Patients With Newly Diagnosed Diabetes: A Randomized Clinical Trial
Brief Title: Metformin and Pioglitazone Effects on Fetuin-A and Osteoprotegrin Concentrations in Type 2 Diabetes Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tehran University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Alireza Esteghamati, Alireza Esteghamati, M.D., Tehran University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 90-111-60037
Record Dates: First submitted 2014-01-02; First posted 2014-01-03 (Estimated); Last update posted 2014-01-03 (Estimated); Status verified 2014-01

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Fetuin-A; OPG; Metformin; Pioglitazone
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Metformin; Pioglitazone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Metformin (Active Comparator): patients receiving fixed dose metformin 1000 mg daily
  Interventions: Drug: Metformin
- Pioglitazone (Active Comparator): patients receiving fixed dose pioglitazone 30 mg daily
  Interventions: Drug: Pioglitazone

INTERVENTIONS:
Drug: Metformin — Metformin 1000 mg fixed dose, twice daily (500 mg tablets x 2)
  Arms: Metformin
Drug: Pioglitazone — Pioglitazone 30 mg fixed dose, twice daily (15 mg tablets x 2)
  Arms: Pioglitazone

SUMMARY:
Oral hypoglycemic agents, along with dietary modification and exercise encompass the mainstay of treatment in early stages of T2DM. Biguanides and thiazolidinediones are two major groups of hypoglycemic medications that while function via different pathways, mare both effective in short- and long-term glucose control. These medications diminish or delay long term micro- and macrovascular complications associated with T2DM although at different rates. Excessive insulin resistance accounts for a sustained increase in cardiovascular incidents in T2DM subjects. Given the shared pathway of insulin resistance/fetuin-A/OPG in atherosclerosis formation, it is conceivable that insulin sensitizing anti-diabetes medications are able to modify successive CAD risk via direct and indirect amelioration of insulin resistance/fetuin-A/OPG. The present study is therefore designed to investigate the effects of metformin and pioglitazone monotherapy on serum concentrations of fetuin-A and OPG in a group of Iranian adults with newly diagnosed T2DM.

ELIGIBILITY:
Inclusion Criteria:

Newly diagnosed type 2 diabetes patients based on American Diabetes Association criteria (2011) for diagnosis of diabetes

Exclusion Criteria:

Previous intake of oral hypoglycemic agents for treatment of diabetes or other hyperglycemia associated conditions Intake of glucocorticoids in the past one year Major illnesses of heart, lung, kidney, and liver.

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2012-01; Primary Completion 2012-03 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Serum concentrations of fetuin-A | 12 weeks
Serum concentrations of osteoprotegrin | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Alireza Esteghamati, M.D, Principal Investigator — Tehran University of Medical Sciences
Locations (1):
- Diabetes Clinic, Vali-Asr Hospital, Tehran University of Medical Sciences, Tehran, Iran

REFERENCES:
- [Derived] Esteghamati A, Afarideh M, Feyzi S, Noshad S, Nakhjavani M. Comparative effects of metformin and pioglitazone on fetuin-A and osteoprotegerin concentrations in patients with newly diagnosed diabetes: A randomized clinical trial. Diabetes Metab Syndr. 2015 Oct-Dec;9(4):258-65. doi: 10.1016/j.dsx.2014.09.009. Epub 2014 Oct 14. PMID 25450818